CLINICAL TRIAL: NCT04472559
Title: Randomized Controlled Trial of Acupressure for Health-Related Quality of Life and Perception of Stress Among Health Care Providers During the COVID-19 Pandemic
Brief Title: Acupressure for COVID-19 Related Quality of Life and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Kakit P. Hui, MD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-000773
Record Dates: First submitted 2020-07-13; First posted 2020-07-15 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Quality of Life; Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-acupressure (Experimental)
  Interventions: Behavioral: Self-acupressure
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Self-acupressure — Self-acupressure
  Arms: Self-acupressure

SUMMARY:
This study is being conducted to evaluate the efficacy of acupressure in promoting health and well-being among healthcare workers during the COVID-19 pandemic. The investigators hypothesize that providing participants with a remote and standardized self-acupressure training program will improve HRQOL and the perception of stress. In the event that the study demonstrates acupressure to be safe and effective for this indication, the training could be scaled up and deployed at low-cost nationally and internationally.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (18 years of age and over) who are health care providers according to self-report will be eligible for participation with the exception of subjects meeting exclusion criteria as below.

Exclusion Criteria:

* Exclusion criteria includes subjects who are physically unable to participate (e.g., from severe arthritis) or cognitively unable to participate (e.g., from dementia) will be excluded. Patients unable to provide their own informed consent will be excluded. Patients under the age of 18 years will be excluded. Pregnant women will be excluded. Patients who have previous training in acupressure will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life | 8 weeks
  SF-12v2
Perception of stress | 8 weeks
  Perceived Stress Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ka-Kit Hui, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abbott R, Hui EK, Kao L, Tse V, Grogan T, Chang BL, Hui KK. Randomized Controlled Trial of Acupressure for Perception of Stress and Health-Related Quality of Life Among Health Care Providers During the COVID-19 Pandemic: The Self-Acupressure for Stress (SAS) Trial. Am J Med Open. 2023 Dec;10:100056. doi: 10.1016/j.ajmo.2023.100056. Epub 2023 Aug 25. PMID 38125337